CLINICAL TRIAL: NCT06273423
Title: A Feasibility Randomized Controlled Evaluation of a Mind-Body Dance Fitness Program for Improving Symptoms of Postpartum Depression
Brief Title: Feasibility Evaluation of a Dance Fitness Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Tracy Hellem, Associate Professor, Montana State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OULA for Postpartum Depression
Record Dates: First submitted 2024-02-08; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Postpartum Depression
Keywords: Postpartum; Depression; Mind-body; Physical activity
MeSH Terms: conditions — Depression, Postpartum; Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group dance fitness, OULA (Experimental): Mind-body dance fitness group
  Interventions: Other: OULA, Mind-body Physical Activity
- Waitlist Control (No Intervention): Waitlist control group

INTERVENTIONS:
Other: OULA, Mind-body Physical Activity — Group dance fitness program with focus on the mind-body connection
  Arms: Group dance fitness, OULA

SUMMARY:
The objective of this pilot project is to assess the feasibility, acceptability, and mental health impact of OULA for women with postpartum depression (PPD).

DETAILED DESCRIPTION:
The proposed project is a pilot two-arm randomized controlled trial (RCT), with specific aims to evaluate the feasibility and acceptability of implementing an RCT of OULA (named after Missoula, MT) for the treatment of postpartum depression, and to explore between-subject changes in postpartum depression and postpartum anxiety following 8-weeks of OULA or waitlist control.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-39 years
* Have an infant 0-12 months old
* Self-report clearance from provider to engage in physical activity following birth
* Structured Clinical Interview for Diagnostic Statistical Manual-5-Research Version (SCID-5-RV) diagnosis of major depressive episode (MDE) with onset during pregnancy or 12 months following childbirth
* Edinburgh Postnatal Depression Scale (EPDS) score of 10 or above
* English speaking
* OULA-naïve
* If on first-line treatment for depression; antidepressant dose must be stable for 6 weeks; psychotherapy duration of treatment must be at least 4 weeks

Exclusion Criteria:

* Unable to be physically active
* Current pregnancy
* SCID-5-RV diagnosis of bipolar disorder, schizophrenia, or current substance use disorder
* Active suicidal attempt or plan identified on the SCID-5-RV
* Suicide attempt in the past 6 months
* Concurrent participation in another group dance fitness format
* No access to Internet via computer, tablet, or smart phone

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability | 7 months
  Feasibility will be evaluated using recruitment, retention, OULA attendance, and treatment completion data, amd intervention fidelity. Feasibility of recruitment will be assessed through the number of participants eligible for randomization, proportion of participants randomized relative to the total number of referrals, and number of participants enrolled each month. Feasibility of intervention will be evaluated through treatment completion and retention rates, Feasibility of Intervention Measure (FIM) will be used at intervention completion. Fidelity assessment will be measured by OULA instructors completing an self-evaluation checklist. Women in the OULA group will complete the 8-item Client Satisfaction Questionnaire (CSQ-8) will be collected at week 8. Acceptability will be assessed through reasons for withdrawal. Acceptability of Intervention Measure (AIM) and Intervention Appropriateness Measure (IAM) will be collected at week 8.

SECONDARY OUTCOMES:
Changes in postpartum depression | 7 months
  The Edinburgh Postnatal Depression Scale will be used at baseline, weeks 4, 8, and 10 to evaluate postpartum depression.
Changes in postpartum anxiety | 7 months
  Postpartum Specific Anxiety Scale Research Short Form will be used at baseline, weeks 4, 8, and 10 to evaluate postpartum anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Hellem, PhD, Principal Investigator — Montana State University

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in mind-body physical activity interventions for postpartum depression. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).